CLINICAL TRIAL: NCT07091344
Title: Evaluation of Cognitive, Metacognitive, Social Cognition and Trauma Related-Variables in Patients With Psychosis Receiving VR-Based Avatar Therapy
Brief Title: Cognitive and Metacognitive Evaluation in VR-Based Avatar Therapy for Psychosis
Acronym: Meta-VR-AVATAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Principal Investigator, Susana Ochoa, PhD, Research Unit Coordinator, Fundació Sant Joan de Déu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-01-24; PS-01-24 (Registry Identifier: ethics comitee Parc Sanitari Sant Joan de Déu)
Record Dates: First submitted 2025-02-11; First posted 2025-07-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia Disorders; Treatment Resistant Hallucinations
Keywords: VR-based Avatar Therapy; cognition; metacognition; social cognition; psychosis; schizophrenia spectrum disorders; auditory hallucinations; trauma and psychosis; emotion recognition; Personalized therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The study employs a single-group pre-post interventional design with a waiting list control phase. All participants will initially undergo a 12-week waiting period (control phase) starting at screening (week 0). Baseline assessments will be conducted at week 12, followed by a 12-week intervention phase where participants receive 7 individual VR-based Avatar Therapy sessions. Post-therapy assessments will be conducted at week 24 to evaluate changes in auditory hallucinations and associated cognitive, metacognitive, and social cognition variables.
  This design allows for a comprehensive evaluation of both the direct effects of the intervention and the potential moderating or mediating role of the measured variables on therapeutic outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VR-Based Avatar Therapy with Cognitive and Metacognitive Assessments (Experimental): Participants will receive VR-based Avatar Therapy over a 12-week intervention period, consisting of 7 individual therapy sessions. This intervention is designed to externalize and reframe distressing auditory hallucinations using virtual reality.
  In addition to the standard therapy, participants will undergo comprehensive assessments of cognition, metacognition, and social cognition at screening (week 0), baseline (week 12), during the intervention (weeks 12-24), and post-therapy (week 24). These measures will evaluate emotional recognition, attributional style, theory of mind, cognitive flexibility, and trauma history, aiming to explore their role in treatment outcomes.
  Interventions: Behavioral: VR-Based Avatar Therapy with Cognitive and Metacognitive Assessments

INTERVENTIONS:
Behavioral: VR-Based Avatar Therapy with Cognitive and Metacognitive Assessments — VR-Based Avatar Therapy is a 12-week intervention designed to help patients with psychosis manage distressing auditory hallucinations. The therapy consists of 7 individual sessions using virtual reality (VR) technology to externalize the auditory hallucinations, allowing patients to interact with a computer-generated avatar representing their dominant voice.
  In addition to standard therapy, participants will undergo assessments of cognition, metacognition, and social cognition to explore their impact on treatment outcomes. These assessments include measures of emotion recognition, attributional style, theory of mind, cognitive flexibility, and trauma history. Sessions are conducted using VR headsets and noise-canceling headphones to enhance immersion, and patients receive ongoing therapeutic guidance throughout the process.

SUMMARY:
This study aims to evaluate the relationship between cognitive, metacognitive and social cognition variables in patients with psychosis undergoing VR-based Avatar Therapy for the treatment of auditory hallucinations. In addition to the primary intervention, participants will be assessed using validated tools for emotion recognition, attributional style, theory of mind, neurocognition, and metacognition. The study also explores the potential role of trauma as a predisposing factor. Assessments will be conducted at four time points: screening (week 0), baseline (week 12), intervention period (weeks 12-24), and post-therapy follow-up (week 24). By investigating these variables, this study seeks to better understand their impact on treatment outcomes and contribute to the development of personalized therapeutic approaches.

DETAILED DESCRIPTION:
This interventional study investigates the impact of cognitive, metacognitive, and social cognition variables on the outcomes of VR-based Avatar Therapy for auditory hallucinations in patients with psychosis. Participants will be assessed at four key time points: screening (week 0), baseline (week 12), during the intervention (weeks 12-24), and post-therapy (week 24).

The intervention consists of 7 individual VR-based Avatar Therapy sessions delivered over 12 weeks. The therapy uses virtual reality to externalize and reframe distressing auditory hallucinations, helping participants develop more adaptive responses.

In addition to evaluating the therapy's effectiveness, the study incorporates validated tools to measure:

Social Cognition: Emotional recognition (Test de Reconocimiento Emocional), attributional style (AIHQ), theory of mind (Hinting Task), and social perception (SFRT-2).

Metacognition: Insight and cognitive monitoring using the BCIS and CBQ. Cognition: Neuropsychological functions, including attention, flexibility, and memory (SCIP, Stroop, TMT, and Vocabulary WAIS).

Trauma as a predisposing factor: Using the Childhood Trauma Questionnaire (CTQ).

By examining these variables, the study aims to deepen the understanding of their influence on treatment outcomes and inform the development of personalized therapeutic approaches for psychosis.

ELIGIBILITY:
**Inclusion Criteria:**

* Adults aged 18 years or older.
* Diagnosis of schizophrenia spectrum disorder according to DSM-5 criteria.
* Experience of persistent auditory hallucinations for at least 3 months (PANSS hallucination score ≥ 3).
* Stable medication dosage for at least 4 weeks prior to recruitment.
* Fluent in the spoken language of the study site (Spanish).
* Able to provide informed consent.
* Regular psychiatric follow-up care.

**Exclusion Criteria:**

* Inability to identify a dominant voice for Avatar Therapy intervention.
* Intellectual disability based on medical history.
* Active substance abuse.
* Central nervous system injury or neurological disorders affecting cognitive performance.
* Severe visual impairment that precludes the use of VR technology.
* Aversion to virtual reality or prior experience of simulator sickness.
* Current suicidal ideation or risk.
* Lack of cooperation or inability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Emotion Recognition Score | Week 0, Week 12, Week 24
  Change in participants' ability to recognize basic emotions using the Faces Test. Score range: 0-20; higher scores = better emotion recognition.
Change in Executive Functioning Score | Week 0, Week 12, Week 24.
  Change in Executive Functioning Score Executive functioning assessed with the Wisconsin Card Sorting Test (WCST). Outcomes include number of categories completed (0-6; higher = better) and number of perseverative errors (no fixed maximum; lower = better). The task ends when the participant completes 6 categories or after all 128 cards are placed.
Change in Attributional Style Score | Week 0, Week 12, Week 24
  Attributional style in ambiguous social situations assessed with the Ambiguous Intentions Hostility Questionnaire (AIHQ). Score range: 0-100; higher scores = greater hostile attribution/conviction.
Change in Theory of Mind Score | Week 0, Week 12, Week 24
  Ability to infer others' intentions measured by the Hinting Task. Score range: 0-6; higher scores = better Theory of Mind.
Change in Metacognition Score | Week 0, Week 12, Week 24
  Cognitive insight measured by the Beck Cognitive Insight Scale (BCIS): Self-reflectiveness (0-27; higher = better) and Self-certainty (0-21; higher = worse).
Change in Cognitive Flexibility Score | Week 0, Week 12, Week 24
  Mental flexibility assessed with the Trail Making Test, Part B. Outcome: time in seconds (maximum 300 seconds); lower times = better performance.
Change in Global Cognitive Performance Score | Week 0, Week 12, Week 24
  Global cognition assessed with the Screen for Cognitive Impairment in Psychiatry (SCIP). Total score range: 0-75; higher = better cognitive performance.
Change in Working Memory Score | Week 0, Week 12, Week 24
  Working memory assessed by the WAIS-IV Digit Span. Scaled score range: 1-19; higher scores = better performance.

OTHER OUTCOMES:
Childhood Trauma Exposure (Baseline moderator) | Week 0 (one-time measure).
  Childhood trauma at baseline measured with the CTQ-SF. Total score range: 25-125; higher = greater trauma exposure.
Change in Verbal Skills Score | Week 0, Week 12, Week 24
  Verbal ability assessed by WAIS-IV Vocabulary. Scaled score range: 1-19; higher scores = better verbal ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Sant Joan de Déu - Unitat de Recerca del Parc Sanitari Sant Joan de Déu, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) will be made available upon reasonable request, after publication of primary results, and subject to approval by the research ethics committee and data protection regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anonymized IPD and supporting documents will be made available after publication of the main study results and for a minimum period of 5 years, starting approximately 12 months after study completion.
Access Criteria: Qualified researchers affiliated with academic or healthcare institutions may request access to anonymized IPD and supporting documents for independent verification or secondary analysis. Requests will be reviewed by the sponsor and must include a data-sharing agreement and ethics approval. Access will be provided through a secure institutional platform.

REFERENCES:
- [Background] Corcoran R, Mercer G, Frith CD. Schizophrenia, symptomatology and social inference: investigating "theory of mind" in people with schizophrenia. Schizophr Res. 1995 Sep;17(1):5-13. doi: 10.1016/0920-9964(95)00024-g. PMID 8541250
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Schmid P, Czekaj A, Frick J, Steinert T, Purdon SE, Uhlmann C. The screen for cognitive impairment in psychiatry (SCIP) as a routinely applied screening tool: pathology of acute psychiatric inpatients and cluster analysis. BMC Psychiatry. 2021 Oct 9;21(1):494. doi: 10.1186/s12888-021-03508-4. PMID 34627191
- [Background] Reitan RM. Trail making test results for normal and brain-damaged children. Percept Mot Skills. 1971 Oct;33(2):575-81. doi: 10.2466/pms.1971.33.2.575. No abstract available. PMID 5124116
- [Background] Beck AT, Baruch E, Balter JM, Steer RA, Warman DM. A new instrument for measuring insight: the Beck Cognitive Insight Scale. Schizophr Res. 2004 Jun 1;68(2-3):319-29. doi: 10.1016/S0920-9964(03)00189-0. PMID 15099613
- [Background] Combs DR, Penn DL, Wicher M, Waldheter E. The Ambiguous Intentions Hostility Questionnaire (AIHQ): a new measure for evaluating hostile social-cognitive biases in paranoia. Cogn Neuropsychiatry. 2007 Mar;12(2):128-43. doi: 10.1080/13546800600787854. PMID 17453895
- [Background] Brebion G, Stephan-Otto C, Cuevas-Esteban J, Usall J, Ochoa S. Impaired memory for temporal context in schizophrenia patients with hallucinations and thought disorganisation. Schizophr Res. 2020 Jun;220:225-231. doi: 10.1016/j.schres.2020.03.014. Epub 2020 Mar 24. PMID 32220501
- [Background] Lorente-Rovira E, Grasa E, Ochoa S, Corripio I, Pelaez T, Lopez-Carrilero R, Gutierrez-Gea A, Morano-Guillen M, Villagran JM, Bartels-Velthuis AA, Jenner JA, Sanjuan J. Different measures for auditory hallucinations in populations with psychosis. The Validation of the Spanish versions of the Auditory Vocal Hallucination Rating Scale (AVHRS) and the Positive and Useful Voices Inquiry (PUVI). Rev Psiquiatr Salud Ment (Engl Ed). 2022 Oct-Dec;15(4):259-271. doi: 10.1016/j.rpsmen.2020.03.002. PMID 36513402
- [Background] Stephan-Otto C, Nunez C, Lombardini F, Cambra-Marti MR, Ochoa S, Senior C, Brebion G. Neurocognitive bases of self-monitoring of inner speech in hallucination prone individuals. Sci Rep. 2023 Apr 17;13(1):6251. doi: 10.1038/s41598-023-32042-4. PMID 37069194
- [Background] Diaz-Cutraro L, Garcia-Mieres H, Dimaggio G, Lysaker P, Moritz S, Ochoa S. Metacognition in psychosis: What and how do we assess it? Span J Psychiatry Ment Health. 2023 Jul-Sep;16(3):206-207. doi: 10.1016/j.rpsm.2022.09.003. Epub 2022 Sep 24. No abstract available. PMID 37716848
- [Background] Garety PA, Edwards CJ, Jafari H, Emsley R, Huckvale M, Rus-Calafell M, Fornells-Ambrojo M, Gumley A, Haddock G, Bucci S, McLeod HJ, McDonnell J, Clancy M, Fitzsimmons M, Ball H, Montague A, Xanidis N, Hardy A, Craig TKJ, Ward T. Digital AVATAR therapy for distressing voices in psychosis: the phase 2/3 AVATAR2 trial. Nat Med. 2024 Dec;30(12):3658-3668. doi: 10.1038/s41591-024-03252-8. Epub 2024 Oct 28. PMID 39468363